CLINICAL TRIAL: NCT01237223
Title: An 8-week Double-blind, Multicenter, Randomized, 6-arm, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of SPA100 (Fixed-dose Combination of Aliskiren and Amlodipine) in Patients With Essential Hypertension
Brief Title: Efficacy and Safety of SPA100 (Fixed-dose Combination of Aliskiren/Amlodipine) in Patients With Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CSPA100A1301
Record Dates: First submitted 2010-10-29; First posted 2010-11-09 (Estimated); Results first posted 2012-06-13 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-05

CONDITIONS: Essential Hypertension
Keywords: Aliskiren; Amlodipine; Essential hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — aliskiren; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo (Placebo Comparator): In order to adequately blind the study, patients were required to take a total of 3 tablets and 2 capsules of study medication throughout the study. In single blind run-in (4 weeks) and double blind treatment period (8 weeks), patients were received matching placebo of aliskiren/amlodipine 150/5 mg tablet, aliskiren/amlodipine 150/2.5 mg tablet, aliskiren 150 mg tablet and two amlodipine 2.5 mg capsules once daily.
  Interventions: Drug: Placebo of Aliskiren; Drug: Placebo of Amlodipine; Drug: Placebo of Aliskiren/amlodipine 150/2.5 mg; Drug: Placebo of Aliskiren/amlodipine 150/5 mg
- Aliskiren 150 mg (Active Comparator): In order to adequately blind the study, patients were required to take a total of 3 tablets and 2 capsules of study medication throughout the study.
  Patients received Aliskiren 150 mg tablet once daily (o.d)+ placebo of two amlodipine 2.5 mg capsule o.d., aliskiren/amlodipine 150/5 mg tablet o.d , aliskiren/amlodipine 150/2.5 mg tablet o.d for 8 weeks of double blind period.
  Interventions: Drug: Aliskiren 150 mg; Drug: Placebo of Amlodipine; Drug: Placebo of Aliskiren/amlodipine 150/2.5 mg; Drug: Placebo of Aliskiren/amlodipine 150/5 mg
- Amlodipine 2.5 mg (Active Comparator): In order to adequately blind the study, patients were required to take a total of 3 tablets and 2 capsules of study medication throughout the study.
  Patients received Amlodipine 2.5 mg capsule once daily (o.d)+ placebo of amlodipine 2.5 mg capsule o.d., Aliskiren 150 mg o.d., aliskiren/amlodipine 150/5 mg tablet o.d , aliskiren/amlodipine 150/2.5 mg tablet o.d for 8 weeks of double blind period.
  Interventions: Drug: Amlodipine 2.5 mg; Drug: Placebo of Aliskiren; Drug: Placebo of Amlodipine; Drug: Placebo of Aliskiren/amlodipine 150/2.5 mg; Drug: Placebo of Aliskiren/amlodipine 150/5 mg
- Amlodipine 5 mg (Active Comparator): In order to adequately blind the study, patients were required to take a total of 3 tablets and 2 capsules of study medication throughout the study.
  Patients received amlodipine 5 mg (two amlodipine 2.5 mg capsules o.d.)+ placebo of aliskiren 150 mg tablet o.d., aliskiren/amlodipine 150/5 mg tablet o.d. , aliskiren/amlodipine 150/2.5 mg tablet o.d. for 8 weeks of double blind period.
  Interventions: Drug: Amlodipine 2.5 mg; Drug: Placebo of Aliskiren; Drug: Placebo of Aliskiren/amlodipine 150/2.5 mg; Drug: Placebo of Aliskiren/amlodipine 150/5 mg
- Aliskiren/amlodipine 150/2.5 mg (Experimental): In order to adequately blind the study, patients were required to take a total of 3 tablets and 2 capsules of study medication throughout the study.
  Patients received aliskiren/amlodipine 150/2.5 mg tablet o.d. + placebo of two amlodipine 2.5 mg capsules o.d., aliskiren 150 mg tablet o.d., aliskiren/amlodipine 150/5 mg tablet o.d. for 8 weeks of double blind period.
  Interventions: Drug: Aliskiren/Amlodipine 150/2.5 mg; Drug: Placebo of Aliskiren; Drug: Placebo of Amlodipine; Drug: Placebo of Aliskiren/amlodipine 150/5 mg
- Aliskiren/amlodipine 150/5 mg (Experimental): In order to adequately blind the study, patients were required to take a total of 3 tablets and 2 capsules of study medication throughout the study.
  Patients received aliskiren/amlodipine 150/5 mg tablet o.d. + placebo of two amlodipine 2.5 mg capsules o.d., aliskiren 150 mg tablet o.d., aliskiren/amlodipine 150/2.5 mg tablet o.d. for 8 weeks of double blind period.
  Interventions: Drug: Aliskiren/amlodipine 150/5 mg; Drug: Placebo of Aliskiren; Drug: Placebo of Amlodipine; Drug: Placebo of Aliskiren/amlodipine 150/2.5 mg

INTERVENTIONS:
Drug: Aliskiren/Amlodipine 150/2.5 mg — Aliskiren/amlodipine 150/2.5 mg tablet
  Arms: Aliskiren/amlodipine 150/2.5 mg
Drug: Aliskiren/amlodipine 150/5 mg — Aliskiren/amlodipine 150/5 mg tablet
  Arms: Aliskiren/amlodipine 150/5 mg
Drug: Aliskiren 150 mg — Aliskiren 150 mg tablet
  Arms: Aliskiren 150 mg
Drug: Amlodipine 2.5 mg — Amlodipine 2.5 mg capsule
  Arms: Amlodipine 2.5 mg; Amlodipine 5 mg
Drug: Placebo of Aliskiren — Aliskiren placebo tablet
  Arms: Aliskiren/amlodipine 150/2.5 mg; Aliskiren/amlodipine 150/5 mg; Amlodipine 2.5 mg; Amlodipine 5 mg; Placebo
Drug: Placebo of Amlodipine — Amlodipine placebo capsule
  Arms: Aliskiren 150 mg; Aliskiren/amlodipine 150/2.5 mg; Aliskiren/amlodipine 150/5 mg; Amlodipine 2.5 mg; Placebo
Drug: Placebo of Aliskiren/amlodipine 150/2.5 mg — Aliskiren/amlodipine 150/2.5 mg placebo tablet
  Arms: Aliskiren 150 mg; Aliskiren/amlodipine 150/5 mg; Amlodipine 2.5 mg; Amlodipine 5 mg; Placebo
Drug: Placebo of Aliskiren/amlodipine 150/5 mg — Aliskiren/amlodipine 150/5 mg placebo tablet
  Arms: Aliskiren 150 mg; Aliskiren/amlodipine 150/2.5 mg; Amlodipine 2.5 mg; Amlodipine 5 mg; Placebo

SUMMARY:
The purpose of the study was to evaluate the efficacy (blood pressure lowering effect) and safety of SPA100 (Fixed-dose Combination of Aliskiren and Amlodipine) in patients with essential hypertension (mean sitting diastolic blood pressure [msDBP] ≥ 95 mmHg and < 110 mmHg and mean sitting systolic blood pressure [msSBP] ≥ 140 mmHg ). This study was conducted to support registration of the fixed-dose combination of aliskiren and amlodipine for the treatment of hypertension in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Patients with essential hypertension (msDBP ≥ 95 mmHg and < 110 mmHg and msSBP ≥140 mmHg )
* Outpatients

Exclusion Criteria:

* Severe hypertension (msDBP ≥110 mmHg and/or msSBP ≥ 180 mmHg)
* History of allergy or hypersensitivity to renin inhibitors, calcium channel blockers
* History or evidence of a secondary hypertension

Other protocol-defined inclusion/exclusion criteria applied

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1342 (Actual)
Dates: Start 2010-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- Japan (11):
  - Investigative Site, Aichi
  - Investigative Site, Ehime
  - Investigative Site, Fukuoka
  - Investigative Site, Hokkaido
  - Investigative Site, Hyōgo
  - Investigative Site, Kanagawa
  - Investigative Site, Kyoto
  - Investigative Site, Okayama
  - Investigative Site, Osaka
  - Investigative Site, Saitama
  - Investigative Site, Tokyo

RESULTS

PARTICIPANT FLOW:
Period: Single Blind(Run-in Period, 4 Weeks)
Arm/Group | Placebo | Aliskiren 150 mg | Amlodipine 2.5 mg | Amlodipine 5 mg | Aliskiren/Amlodipine 150/2.5 mg | Aliskiren/Amlodipine 150/5 mg
Started | 1342 (All the patients enrolled to single blind period received only placebo treatment.) | 0 | 0 | 0 | 0 | 0
Completed | 944 | 0 | 0 | 0 | 0 | 0
Not Completed | 398 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 29 | 0 | 0 | 0 | 0 | 0
Not completed — Abnormal laboratory value(s) | 25 | 0 | 0 | 0 | 0 | 0
Not completed — Abnormal test procedure result(s) | 308 | 0 | 0 | 0 | 0 | 0
Not completed — Subject withdrew consent | 28 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol deviation(s) | 8 | 0 | 0 | 0 | 0 | 0
Period: Double Blind (Treatment Period, 8 Weeks)
Arm/Group | Placebo | Aliskiren 150 mg | Amlodipine 2.5 mg | Amlodipine 5 mg | Aliskiren/Amlodipine 150/2.5 mg | Aliskiren/Amlodipine 150/5 mg
Started | 153 | 157 | 158 | 158 | 159 | 159
Completed | 120 | 142 | 143 | 153 | 155 | 154
Not Completed | 33 | 15 | 15 | 5 | 4 | 5
Not completed — Adverse Event | 12 | 4 | 3 | 2 | 2 | 1
Not completed — Unsatisfactory therapeutic effect | 20 | 6 | 7 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 4 | 4 | 0 | 1 | 1
Not completed — Administrative problems | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol deviation(s) | 0 | 1 | 1 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: In order to adequately blind the study, patients were required to take a total of 3 tablets and 2 capsules of study medication throughout the study. Patients were received matching placebo of aliskiren/amlodipine 150/5 mg tablet, aliskiren/amlodipine 150/2.5 mg tablet, aliskiren 150 mg tablet and two amlodipine 2.5 mg capsules once daily for 8 weeks of double blind period.
- Total: Total of all reporting groups
Arm/Group | Placebo | Aliskiren 150 mg | Amlodipine 2.5 mg | Amlodipine 5 mg | Aliskiren/Amlodipine 150/2.5 mg | Aliskiren/Amlodipine 150/5 mg | Total
Number analyzed (Participants) | 153 | 157 | 158 | 158 | 159 | 159 | 944
Age Continuous [Mean (Standard Deviation); unit: years] — Baseline measurements were based on randomized patients.
  years | 54.6 (8.35) | 55.0 (9.96) | 54.8 (10.25) | 55.8 (10.05) | 54.6 (11.11) | 55.5 (9.86) | 55.1 (9.96)
Age, Customized [Number; unit: participants]
  < 65 years | 128 | 131 | 129 | 126 | 125 | 127 | 766
  >=65 years | 25 | 26 | 29 | 32 | 34 | 32 | 178
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 39 | 45 | 51 | 51 | 57 | 288
  Male | 108 | 118 | 113 | 107 | 108 | 102 | 656

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (msDBP) to End of Study (Week 8)
Description: Sitting blood pressure was measured at trough (24 hours ± 2 hours post dose) and recorded at all study visits. At the first study visit, blood pressure was measured in both arms and the arm with highest sitting DBP was found and used for all subsequent readings throughout the study. The repeat sitting measurements were made at 1-2 minute intervals and the mean of these three sitting blood pressure measurements were used as the average sitting blood pressure for that visit. Analysis of covariance (ANCOVA) model contained treatment and region as two factors and baseline as a covariate.
Time Frame: Baseline, Week 8
Population: Full analysis set (FAS): All randomized patients received at least one dose of double-blind study medication.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Groups:
- Placebo: In order to adequately blind the study, patients were required to take a total of 3 tablets and 2 capsules of study medication throughout the study. Patients were received matching placebo of aliskiren/amlodipine 150/5 mg tablet, aliskiren/amlodipine 150/2.5 mg tablet, aliskiren 150 mg tablet and two amlodipine 2.5 mg capsules once daily for 8 weeks of double blind treatment period.
Arm/Group | Placebo | Aliskiren 150 mg | Amlodipine 2.5 mg | Amlodipine 5 mg | Aliskiren/Amlodipine 150/2.5 mg | Aliskiren/Amlodipine 150/5 mg
Number analyzed (Participants) | 153 | 157 | 158 | 158 | 159 | 159
mm Hg | -5.21 (0.69) | -7.49 (0.68) | -9.46 (0.68) | -11.90 (0.68) | -12.40 (0.68) | -16.43 (0.68)

2. Secondary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP) to End of Study (Week 8)
Description: as for outcome 1
Time Frame: Baseline, Week 8
Population: Full analysis set (FAS): All randomized patients received at least one dose of double-blind study medication.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo | Aliskiren 150 mg | Amlodipine 2.5 mg | Amlodipine 5 mg | Aliskiren/Amlodipine 150/2.5 mg | Aliskiren/Amlodipine 150/5 mg
Number analyzed (Participants) | 153 | 157 | 158 | 158 | 159 | 159
mm Hg | -4.57 (0.97) | -10.63 (0.96) | -13.16 (0.96) | -17.98 (0.96) | -18.15 (0.96) | -25.49 (0.96)

3. Secondary Outcome: Percentage of Participants Achieving Blood Pressure Control at Endpoint
Description: Blood pressure control is defined as having as a msDBP < 90 mmHg and a msSBP < 140 mmHg.
Time Frame: 8 weeks
Population: Full analysis set (FAS) included all randomized patients received at least one dose of double-blind study medication
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Aliskiren 150 mg | Amlodipine 2.5 mg | Amlodipine 5 mg | Aliskiren/Amlodipine 150/2.5 mg | Aliskiren/Amlodipine 150/5 mg
Number analyzed (Participants) | 153 | 157 | 158 | 158 | 159 | 159
percentage of participants | 16.3 | 25.5 | 32.9 | 50.0 | 45.9 | 69.2

4. Secondary Outcome: Percentage of Participants Achieving a Successful Response Rate
Description: The response rate was defined as percentage of participants who achieved msDBP < 90 mmHg or its reduction ≥ 10 mmHg from baseline to endpoint.
Time Frame: 8 weeks
Population: Full analysis set (FAS) included all randomized patients received at least one dose of double-blind study medication
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Aliskiren 150 mg | Amlodipine 2.5 mg | Amlodipine 5 mg | Aliskiren/Amlodipine 150/2.5 mg | Aliskiren/Amlodipine 150/5 mg
Number analyzed (Participants) | 153 | 157 | 158 | 158 | 159 | 159
percentage of participants | 34.6 | 46.5 | 50.6 | 70.3 | 65.4 | 86.2

5. Secondary Outcome: Number of Participants With Adverse Events, Serious Adverse Events and Death
Description: Number of patients with adverse events regardless of study drug relationship during the double-blind treatment period were reported. Serious adverse events of double blind period were reported.
Time Frame: 8 weeks
Population: Safety set: All patients who received at least one dose of double-blind study medication.
Measure: Number; unit: Participants
Arm/Group | Placebo | Aliskiren 150 mg | Amlodipine 2.5 mg | Amlodipine 5 mg | Aliskiren/Amlodipine 150/2.5 mg | Aliskiren/Amlodipine 150/5 mg
Number analyzed (Participants) | 153 | 157 | 158 | 158 | 159 | 159
Participants
  Adverse Events | 62 | 57 | 50 | 49 | 57 | 59
  Serious Adverse Events | 0 | 0 | 2 | 1 | 0 | 1
  Death | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Placebo (Double Blind): In order to adequately blind the study,patients were required to take a total of 3 tablets and 2 capsules of study medication throughout the study. In double blind treatment period (8 weeks), patients were received matching placebo of aliskiren/amlodipine 150/5 mg tablet, aliskiren/amlodipine 150/2.5 mg tablet, aliskiren 150 mg tablet and two amlodipine 2.5 mg capsules once daily.
- Placebo (Single-Blind run-in Period): In order to adequately blind the study,patients were required to take a total of 3 tablets and 2 capsules of study medication throughout the study. In single blind run-in period (4 weeks), patients were received matching placebo of aliskiren/amlodipine 150/5 mg tablet, aliskiren/amlodipine 150/2.5 mg tablet, aliskiren 150 mg tablet and two amlodipine 2.5 mg capsules once daily.
Arm/Group | Placebo (Double Blind) | Aliskiren 150 mg | Amlodipine 2.5 mg | Amlodipine 5 mg | Aliskiren/Amlodipine 150/2.5 mg | Aliskiren/Amlodipine 150/5 mg | Placebo (Single-Blind run-in Period)
Serious Adverse Events (participants affected / at risk) | 0/153 | 0/157 | 2/158 | 1/158 | 0/159 | 1/159 | 4/1342
Other Adverse Events (participants affected / at risk) | 21/153 | 21/157 | 17/158 | 21/158 | 17/159 | 19/159 | 136/1342
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Double Blind) (N=153) | Aliskiren 150 mg (N=157) | Amlodipine 2.5 mg (N=158) | Amlodipine 5 mg (N=158) | Aliskiren/Amlodipine 150/2.5 mg (N=159) | Aliskiren/Amlodipine 150/5 mg (N=159) | Placebo (Single-Blind run-in Period) (N=1342)
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes zoster oticus (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertensive encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Putamen haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Double Blind) (N=153) | Aliskiren 150 mg (N=157) | Amlodipine 2.5 mg (N=158) | Amlodipine 5 mg (N=158) | Aliskiren/Amlodipine 150/2.5 mg (N=159) | Aliskiren/Amlodipine 150/5 mg (N=159) | Placebo (Single-Blind run-in Period) (N=1342)
Nasopharyngitis (Infections and infestations) | 11 | 17 | 14 | 19 | 16 | 16 | 81
Headache (Nervous system disorders) | 12 | 5 | 3 | 2 | 1 | 3 | 59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.